CLINICAL TRIAL: NCT05178420
Title: Discontinuing Statins in Multimorbid Older Adults Without Cardiovascular Disease (STREAM) - a Randomized Non-inferiority Clinical Trial
Brief Title: STREAM Trial - Statins in Multimorbid Older Adults Without Cardiovascular Disease
Acronym: STREAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STREAM
Record Dates: First submitted 2021-11-15; First posted 2022-01-05 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Statin Treatment for Primary Prevention
Keywords: Multimorbidity; Primary prevention; Older adults; Deprescribing; Statin

STUDY DESIGN:
Intervention Model Description: Study subjects are randomly assigned in a 1:1 ratio to either discontinue (intervention arm) or continue (control arm) statin therapy
Who Masked: Outcomes Assessor
Masking Description: The study is open-label, with blinded outcome adjudication. Identification of potential outcome events is performed by blinded study team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin discontinuation (Experimental): Discontinuation of statin therapy - statin therapy will be stopped from the next scheduled intake after study inclusion (intervention arm).
  Interventions: Other: Statin discontinuation
- Statin continuation (No Intervention): Continuation of statin therapy - no change in the prescribed statin therapy (control arm).

INTERVENTIONS:
Other: Statin discontinuation — Statin therapy will be stopped. Additional lipid-lowering medication lowering LDL cholesterol will also be stopped.
  Other Names: Intervention arm
  Arms: Statin discontinuation

SUMMARY:
Statins are among the most widely used drugs. While they were found to be effective for primary and secondary prevention of cardiovascular disease (CVD) in middle-aged subjects, their benefits for primary prevention in older adults (aged ≥70 years) without CVD are uncertain, particularly for those with multimorbidity. The aim of this randomized controlled trial (RCT) is to provide guidance on the benefits and risks of statin deprescribing in multimorbid older adults.

DETAILED DESCRIPTION:
Background:

Until now, no RCT examining the benefits of statins in primary prevention has exclusively recruited multimorbid participants aged 70 years and older (70+), and 70+ participants are under-represented in most RCTs, including those examining statin benefits for primary prevention. However, statin side effects and drug interactions are common in populations of multimorbid older adults and might negatively impact quality of life. The proportion of patients developing myalgia on statins has been shown to be as high as 5-20% in observational studies; older age and polypharmacy are known risk factors for developing muscle problems under statins. Furthermore, multimorbid older adults with polypharmacy are more likely to experience side effects with statins (e.g. elevated liver enzymes, diabetes, myopathy, rhabdomyolysis) and drug-drug interactions (e.g. antibiotics, antifungals), with the potential consequences of drug toxicity, reduced physical activity, sarcopenia and falls. In practice, statins are often discontinued in multimorbid older adults without CVD after side effects. The net clinical benefit of statins for primary prevention in multimorbid 70+ older adults remains unclear, and the effect of multimorbidity might shift the evidence towards favoring no statin treatment, but no large RCT examined this issue.

Design:

The study is a multicenter, randomized, non-inferiority trial conducted in multiple centers in Switzerland, France and the Netherlands. Study subjects are randomly assigned in a 1:1 ratio to either discontinue (intervention arm) or continue (control arm) statin therapy. The study is open-label, with blinded outcome adjudication. After inclusion the study participants will be followed with phone calls, first after 3 months and then yearly for a mean of 24 months (min. follow-up period 12 months, max. follow-up period 48 months). Outcomes are assessed at each study follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥70 years of age
* Multimorbid with ≥2 coexistent chronic conditions (defined by ICD-10 codes) with an estimated duration of 6 months or more based on clinical decision, besides dyslipidemia treated by statins
* Intake of a statin for ≥80% of the time during the year before enrollment

Exclusion Criteria:

1. Cardiovascular secondary prevention setting based on previous large statin trials, defined as:

   * History of myocardial infarction type 1 (NSTEMI/STEMI), OR
   * History of unstable angina, defined as ACS symptomatic at rest, crescendo or new-onset angina (CCS 2 or 3) without ECG or cardiac biomarker changes (based on available documents), OR
   * Stable angina pectoris with a documented ischemia on a stress test or with a significant coronary disease defined as a coronary stenosis >50%, OR
   * History of percutaneous coronary intervention (balloon or stent) or coronary artery bypass graft, OR
   * History of Stroke (does not apply to clearly cardio-embolic causes for stroke e.g. due to atrial fibrillation), OR
   * History of Transient Ischemic Attack, defined as transient neurological deficit without diffusion restriction in MRI, OR
   * History of carotid revascularization (stent, bypass, CEA (carotid thrombendartectomy)), OR
   * History of peripheral arterial disease requiring revascularization (e.g. PTA (percutaneous transluminal angioplasty), stent, femoral TEA (thrombendartectomy), bypass; Fontaine IV)
2. Aortic disease that required a vascular repair or aortic aneurysm with a maximum diameter >5.5 cm (men) or >5.2 cm (women) based on available documents
3. Diagnosis of familial hypercholesterolemia based on Dutch lipid score ≥6 based on available documents (LDL cholesterol, family history, personal history)
4. Elevated risk of death within 3 months after baseline, defined as:

   * Hospitalized patients planned for palliative care within 24h of admission OR
   * Hospitalized patients with a Palliative Performance Scale (PPS) level <30% (based on situation at least 1 month before hospitalization), this corresponds to an estimated survival of 43% after 3 months; OR
   * Patients with an advanced metastatic cancer prognosis of ≤20% survival rate within 1 year after baseline (based on: https://cancersurvivalrates.com)
5. Participation to a clinical trial with potential impact on the STREAM cardiovascular endpoints (based on clinical judgment)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1881 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause death and major non-fatal CV events (non-fatal myocardial infarction, non-fatal ischemic stroke) | 24 months
  The primary endpoint is a composite endpoint of all-cause death and major non-fatal CV events (non-fatal myocardial infarction, non-fatal ischemic stroke). All-cause death (and not CV death only) is chosen to account for a possible shift from CV to other causes of death. The composite endpoint was selected to assess the net clinical benefit in this population with expected high mortality. The clinical event committee which classifies suspected events for the primary and secondary clinical outcomes is blinded. The primary analysis timeframe is at 24 months, and data collection is performed up to 48 months.

SECONDARY OUTCOMES:
Composite endpoint of all-cause death and major non-fatal CV events (non-fatal myocardial infarction, non-fatal ischemic stroke) | up to 48 months
  Composite endpoint of all-cause death and major non-fatal CV events (non-fatal myocardial infarction, non-fatal ischemic stroke).
All-cause death | up to 48 months
  All deaths (for any reason)
Non-CV death | up to 48 months
  All deaths except of deaths due to major CV events
Major CV events | up to 48 months
  CV death, non-fatal myocardial infarction and non-fatal ischemic stroke
Total CV events | up to 48 months
  CV death, non-fatal myocardial infarction, hospitalization for unstable angina, non-fatal ischemic stroke (including TIA) and arterial revascularization (coronary and peripheral urgent and non-urgent revascularization)
Total composite events | up to 48 months
  All-cause death, non-fatal myocardial infarction, hospitalization for unstable angina, non-fatal ischemic stroke (including TIA) and arterial revascularization (coronary and peripheral urgent and non-urgent revascularization)
EQ-5D questionnaire | 3, 12 (primary analysis), 24, 36, 48 months
  EQ-5D is the name of the instrument and not an acronym. General quality of life assessment. The possible range of scores goes from 0 to 1.0, with higher scores indicating better quality of life.
Verbal numeric pain rating score (VNPRS) | 3 months
  To assess statin associated muscle symptoms. The VNPRS is an 11-point scale scored from 0-10, with higher scores indicating higher degree of pain.
Self-reported falls | 12 months
  Self-reported falls, each participant will collect and list all falls during the first 12 months after randomization. Circumstances and medical consequences of each fall will be collected. Aggregated as rate of falls (falls per person per year).
Strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F questionnaire) | 12 (primary analysis), 24, 36, 48 months
  5-item questionnaire, the score ranges from 0 to 10 with higher scores indicating higher degree of sarcopenia.
Girerd medication adherence scale | 12 (primary analysis), 24, 36, 48 months
  6-item questionnaire, the score ranges from 0 to 6, higher scores indicating worse medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD, MAS, Principal Investigator — University of Bern
Locations (24):
- UNIVERSITY HOSPITAL CENTER of Bordeaux, Bordeaux, Nouvelle Acquitaine, France
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands
- Switzerland (22):
  - Klinik Barmelweid AG, Barmelweid, Canton of Aargau
  - Centre hospitalier Bienne, Biel/Bienne, Canton of Bern
  - Spital Limmattal, Schlieren, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Luzerner Höhenklinik Montana AG, Crans-Montana, Valais
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Clinic for General Internal Medicine, Bern University Hospital Bern, Bern
  - Hospital Burgdorf, Burgdorf
  - HFR Fribourg, Fribourg
  - Hôpital La Tour, Geneva
  - Hôpitaux Universitaires de Genève (Geriatrics), Geneva
  - Hôpitaux Universitaires de Genève (Internal Medicine), Geneva
  - Hospital Langnau, Langnau
  - CHUV Lausanne, Lausanne
  - Hôpital Neuchâtelois, Neuchâtel
  - Hospital St. Gallen (Geriatrics), Sankt Gallen
  - Kantonsspital Schaffhausen, Schaffhausen
  - Stadspital Waid, Zurich
  - Stadtspital Triemli, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in the BORIS Research Data, the research data repository of the University of Bern. BORIS Research Data allows searching and is indexed by search engines. All items are stored with a unique Digital Object Identifier (DOI) that can be referenced in respective publication. It should be noted that the investigators plan to register and deposit data that relates to individual, primary publications and not the whole study database as such, as the investigators will use them for secondary analysis. This enables other researchers to replicate published analyses and results as well as to re-use the data for additional analyses such as metaanalysis.
  It is planned to disseminate the results of the trial to key target groups using the Lavis' framework for research knowledge transfer
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Foreseen for one year after publication of the main trial results. Items will be retained indefinitely.
Access Criteria: All efforts will be made to protect privacy and to de-identify the data. However, datasets contain sensitive data. Therefore, data will be shared on request under the following conditions:
  * A meaningful study question by the requester
  * Outline of the planned analyses
  * Valid methodology Signed data sharing agreement that contains a confidentiality agreement and other obligations to ensure privacy of trial participants
URL: https://boris.unibe.ch/policies.html

REFERENCES:
- [Background] Byrne P, Cullinan J, Smith SM. Statins for primary prevention of cardiovascular disease. BMJ. 2019 Oct 16;367:l5674. doi: 10.1136/bmj.l5674. No abstract available. PMID 31619406
- [Background] Shepherd J, Blauw GJ, Murphy MB, Bollen EL, Buckley BM, Cobbe SM, Ford I, Gaw A, Hyland M, Jukema JW, Kamper AM, Macfarlane PW, Meinders AE, Norrie J, Packard CJ, Perry IJ, Stott DJ, Sweeney BJ, Twomey C, Westendorp RG; PROSPER study group. PROspective Study of Pravastatin in the Elderly at Risk. Pravastatin in elderly individuals at risk of vascular disease (PROSPER): a randomised controlled trial. Lancet. 2002 Nov 23;360(9346):1623-30. doi: 10.1016/s0140-6736(02)11600-x. PMID 12457784
- [Background] Han BH, Sutin D, Williamson JD, Davis BR, Piller LB, Pervin H, Pressel SL, Blaum CS; ALLHAT Collaborative Research Group. Effect of Statin Treatment vs Usual Care on Primary Cardiovascular Prevention Among Older Adults: The ALLHAT-LLT Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):955-965. doi: 10.1001/jamainternmed.2017.1442. PMID 28531241
- [Background] Cholesterol Treatment Trialists' Collaboration. Efficacy and safety of statin therapy in older people: a meta-analysis of individual participant data from 28 randomised controlled trials. Lancet. 2019 Feb 2;393(10170):407-415. doi: 10.1016/S0140-6736(18)31942-1. PMID 30712900
- [Background] Ruscica M, Macchi C, Pavanello C, Corsini A, Sahebkar A, Sirtori CR. Appropriateness of statin prescription in the elderly. Eur J Intern Med. 2018 Apr;50:33-40. doi: 10.1016/j.ejim.2017.12.011. Epub 2018 Jan 5. PMID 29310996
- [Background] van der Ploeg MA, Streit S, Achterberg WP, Beers E, Bohnen AM, Burman RA, Collins C, Franco FG, Gerasimovska-Kitanovska B, Gintere S, Gomez Bravo R, Hoffmann K, Iftode C, Pestic SK, Koskela TH, Kurpas D, Maisonneuve H, Mallen CD, Merlo C, Mueller Y, Muth C, Petrazzuoli F, Rodondi N, Rosemann T, Sattler M, Schermer T, Ster MP, Svadlenkova Z, Tatsioni A, Thulesius H, Tkachenko V, Torzsa P, Tsopra R, Tuz C, Vaes B, Viegas RPA, Vinker S, Wallis KA, Zeller A, Gussekloo J, Poortvliet RKE. Patient Characteristics and General Practitioners' Advice to Stop Statins in Oldest-Old Patients: a Survey Study Across 30 Countries. J Gen Intern Med. 2019 Sep;34(9):1751-1757. doi: 10.1007/s11606-018-4795-x. Epub 2019 Jan 16. PMID 30652277
- [Background] Kutner JS, Blatchford PJ, Taylor DH Jr, Ritchie CS, Bull JH, Fairclough DL, Hanson LC, LeBlanc TW, Samsa GP, Wolf S, Aziz NM, Currow DC, Ferrell B, Wagner-Johnston N, Zafar SY, Cleary JF, Dev S, Goode PS, Kamal AH, Kassner C, Kvale EA, McCallum JG, Ogunseitan AB, Pantilat SZ, Portenoy RK, Prince-Paul M, Sloan JA, Swetz KM, Von Gunten CF, Abernethy AP. Safety and benefit of discontinuing statin therapy in the setting of advanced, life-limiting illness: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):691-700. doi: 10.1001/jamainternmed.2015.0289. PMID 25798575
- [Derived] Aebi PS, Adam L, Haller M, Bardoczi JB, Gencer B, Bonnet F, Beer JH, Carballo S, Christ-Crain M, Feller M, Gabutti L, Haynes AG, Moutzouri E, Chocano-Bedoya PO, Bassetti S, Escher R, Egger M, Poortvliet RKE, Schuetz P, Trelle S, Wertli MM, Zekry D, Mean M, Aujesky D, Bauer D, Blum MR, Rodondi N. Rationale and design of 'discontinuing statins in multimorbid older adults without cardiovascular disease (STREAM)': study protocol of a randomised non-inferiority clinical trial. BMJ Open. 2025 May 23;15(5):e093833. doi: 10.1136/bmjopen-2024-093833. PMID 40409969